CLINICAL TRIAL: NCT00612690
Title: Mental Health Services & Predictors of Learning in Urban Schools
Brief Title: School-Based Mental Health Services for Urban Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marc Atkins, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH073749 (NIH); R01MH073749 (NIH); DSIR 82-SECHC (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-12 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Conduct Disorder; Oppositional Defiant Disorder; Attention Deficit Disorder With Hyperactivity
Keywords: Children; School-Based Mental Health Services; Urban Poverty
MeSH Terms: conditions — Conduct Disorder; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Links to Learning (Experimental): Participants received the community mental health consultation model program.
  Interventions: Behavioral: Community mental health consultation model program
- Services as Usual (Active Comparator): Participants received treatment as usual and referrals.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Community mental health consultation model program — The community mental health consultation model program included collaboration among community mental health providers and (1) parent advocates to effectively maintain families in a school-based mental health program, (2) classroom teachers to enhance children's academic performance, and (3) peer-identified influential teachers to influence classroom teachers' use of behavior management strategies. This model further focused on the strongest teacher and parent predictors of student learning.
  Other Names: Links to Learning (L2L)
  Arms: Links to Learning
Behavioral: Treatment as usual (TAU) — TAU included referral to community mental health clinic-based services, where participants received standard care for mental health-related problems.
  Arms: Services as Usual

SUMMARY:
This study will evaluate the effectiveness of school- and home-based mental health services and training modules in supporting learning and behavior in financially disadvantaged children who live in urban areas.

DETAILED DESCRIPTION:
There are an estimated 4.5 to 6.3 million children with mental disorders in the United States. Emotional and behavioral problems associated with childhood mental disorders have a significant impact, with affected children at an increased risk of reduced quality of life and school dropout. If left untreated, childhood mental disorders may continue into adulthood, often impairing ability to function as an adult. It is believed that, compared to clinic-based services, school- and home-based mental health services may lead to greater improvements in children's learning and behavior at school and home. Especially important to this type of approach is a collaborative effort among parents, teachers, and children to encourage and maintain positive behaviors and academic performance both at home and in the classroom. This study evaluated the effectiveness of school- and home-based mental health services and training modules in supporting learning and behavior in financially disadvantaged children who live in urban areas.

This 3-year study involved parent, child, and teacher participants. During Year 1, teacher participants attended a professional development series that focused on strategies that classroom teachers can use to help children with learning and behavior problems at school. The series involved weekly 30-minute sessions, which were held before and after school hours, for a total of 6 months. Teachers completed a brief survey about the content and structure of sessions at the end of each session and gave a monthly review on how they applied their new strategies in the classroom setting. Teachers continued to attend booster sessions of up to 1 hour each month during Year 2. Teachers also participated in periodic case consultation meetings with parents and mental health providers to further develop ways to improve student participants' learning and behavior.

Child participants received either the community mental health program associated with their school or received general clinic-based services (Treatment as usual). The school component of the mental health program consisted of a classroom environment in which the teachers implemented their newly learned strategies to enhance the academic and behavioral performance of the child participants. Parents of child participants in the community mental health program were invited to attend a series of parent/teacher meetings and home visits where mental health service providers discussed strategies that parents and teachers can use to help improve their children's learning and behavior. Parents completed a brief questionnaire at the end of each meeting and gave a monthly review of how they implemented their new strategies in the home setting. Parents continued to communicate with research staff regarding services provided throughout the study.

Assessments for all participants occurred five times over 3 years. Assessments for parent participants included questions about their child's behavior at school and home, their child's use of mental health services, involvement in their child's schooling, and possible stresses in life. Assessments for teachers included questions about the behavior and academic performances of the child participants, parent involvement with the children's schooling, and stresses in their work environment. A research staff member also conducted a 2-hour classroom observation five times over 3 years. Individual child participants were also observed in the classroom by research staff for three 15-minute intervals five times over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Student in kindergarten through 4th grade in a participating school
* Diagnosis of conduct disorder, oppositional defiant disorder, or attention deficit hyperactivity disorder as confirmed by parent and/or teacher report
* Parents and teachers of these students were also eligible to participate

Exclusion Criteria:

* Severe developmental or medical disability

Note: Teachers, parents, and mental health providers of the children enrolled in the study were also consented as per directions from our Institutional Review Board (IRB) because we were asking about sensitive information. Therefore, the ages listed below are for the children enrolled in the study as this was the determining criteria for study participation. Ages of participating adults (i.e., parents and teachers) were included in Baseline Characteristics to provide a complete description of the study participants. However, although adults participated in the study, the eligibility criteria were based on child characteristics as noted above.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 482 (Actual)
Dates: Start 2005-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S. Atkins, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Institute for Juvenile Research, Chicago, Illinois, United States

REFERENCES:
- [Background] Mehta TG, Atkins MS, Frazier SL. The Organizational Health of Urban Elementary Schools: School Health and Teacher Functioning. School Ment Health. 2013 Sep 1;5(3):144-154. doi: 10.1007/s12310-012-9099-4. PMID 23935763
- [Background] Neal JW, Neal ZP, Atkins MS, Henry DB, Frazier SL. Channels of change: contrasting network mechanisms in the use of interventions. Am J Community Psychol. 2011 Jun;47(3-4):277-86. doi: 10.1007/s10464-010-9403-0. PMID 21181552
- [Background] Neal, JW, Shernoff, ES, Frazier, S.L, Stachowicz, E, Frangos, U, & Atkins, MS (2008). Change from within: Engaging teacher key opinion leaders in the diffusion of interventions in urban schools. The Community Psychologist, 41:2, 53-57
- [Background] Atkins MS, Frazier SL. Expanding the Toolkit or Changing the Paradigm: Are We Ready for a Public Health Approach to Mental Health? Perspect Psychol Sci. 2011 Sep;6(5):483-7. doi: 10.1177/1745691611416996. PMID 26168200
- [Background] Atkins MS, Hoagwood KE, Kutash K, Seidman E. Toward the integration of education and mental health in schools. Adm Policy Ment Health. 2010 Mar;37(1-2):40-7. doi: 10.1007/s10488-010-0299-7. PMID 20309623

RESULTS

PARTICIPANT FLOW:
Groups:
- Links to Learning: Participants underwent the community mental health consultation model program.
  Community mental health consultation model program : The community mental health consultation model program included collaboration among community mental health providers and (1) parent advocates to effectively maintain families in a school-based mental health program, (2) classroom teachers to enhance children's academic performance, and (3) peer-identified influential teachers to influence classroom teachers' use of behavior management strategies. This model further focused on the strongest teacher and parent predictors of student learning.
- Services as Usual: Participants received treatment as usual and referrals.
  Treatment as usual (TAU) : TAU included referral to community mental health clinic-based services, where participants received standard care for mental health-related problems.
Period: Overall Study
Arm/Group | Links to Learning | Services as Usual
Started | 275 | 207
Completed | 160 | 89
Not Completed | 115 | 118
Not completed — Lost to Follow-up | 72 | 98
Not completed — Withdrawal by Subject | 32 | 20
Not completed — Withdrawal by Site | 11 | 0

BASELINE CHARACTERISTICS:
Population: Total number of students, teachers, parents, and service providers (in the Links to Learn condition only) who were consented to participate in the study (Note: Service providers in the Services as Usual condition were not research participants).
Groups:
- Links to Learning: Mental health intervention focused on enhancing the predictors of young children's school success
- Services As Usual: Referral to nearby community mental heath agencies for clinic-based services where participants received standard care for mental health-related problems.
- Total: Total of all reporting groups
Arm/Group | Links to Learning | Services As Usual | Total
Number analyzed (Participants) | 289 | 193 | 482
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 104 | 67 | 171
  Between 18 and 65 years | 185 | 126 | 311
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Students | 7.42 (1.81) | 7.66 (1.53) | 7.51 (1.71)
  Teachers | 41.44 (13.46) | 35.58 (11.46) | 38.37 (12.73)
  Service Providers | 32.46 (8.73) | NA (NA) — Service providers in this condition were not research participants. | 32.46 (8.73)
  Parents | 32.06 (7.92) | 32.64 (8.44) | 32.28 (8.10)
Sex/Gender, Customized [Number; unit: participants]
  Students: Male | 74 | 50 | 124
  Students: Female | 30 | 17 | 47
  Teachers: Male | 9 | 7 | 16
  Teachers: Female | 62 | 58 | 120
  Service Provders: Male | 4 | NA — Service providers in this condition were not research participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Service Providers: Female | 13 | NA — Service providers in this condition were not research participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Parents: Male | 1 | 6 | 7
  Parents: Female | 96 | 55 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 130 | 331
  Male | 88 | 63 | 151
Region of Enrollment [Number; unit: participants]
  United States | 289 | 193 | 482

OUTCOME MEASURES:

1. Primary Outcome: Social Skills Rating System (Parent Report)
Description: This rating scale was completed by parents to assess how frequently their child engaged in a range of disruptive, prosocial, and academic behaviors (0 = Never to 2 = Very Often). Normative data are provided by age and sex and the measure was standardized on a heterogeneous population of which one third were urban and 28% were minorities. The scale score, Social Skills, was the primary outcome measure. Scores are rated on a scale of 0 (Never) to 2 (Very Often). The scale score, Social Skills, containing 38 items, was the primary outcome measure. Scores range from 0 to 76 with higher scores indicating improved social skills.
Time Frame: Measured at pre- and post-school year for 3 years
Population: Child participants with available data were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Services as Usual: Participants received treatment as usual and referrals.
  Treatment as usual (TAU) : TAU included referral to community mental health clinic-based services where participants received standard care for mental health-related problems.
Arm/Group | Links to Learning | Services as Usual
Number analyzed (Participants) | 104 | 67
units on a scale
  Baseline | 46.37 (11.97) | 43.25 (10.98)
  Spring Year 1 | 45.02 (10.65) | 41.66 (10.79)
  Fall Year 2 | 47.53 (13.13) | 42.53 (11.45)
  Spring Year 2 | 47.54 (12.24) | 44.63 (9.64)
  Fall Year 3 | 46.95 (13.03) | 38.56 (6.70)
  Spring Year 3 | 48.35 (11.61) | 40.55 (11.22)

2. Secondary Outcome: The Academic Competence Evaluation Scale (ACES)
Description: The ACES is a teacher rating scale that describes a set of behaviors and attitudes measuring teachers' perceptions of student's academic competence and performance. The scale consists of 30 items rated on a 5-point scale (1 = Never, 2 = Seldom, 3 = Sometimes, 4 = Often, 5 = Almost Always). The total score was reported as a mean per item with higher scores indicating better academic competence. Scores could range from 1 to 30.
Time Frame: Measured at pre- and post-school year for 3 years
Population: Only children with available data were included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Links to Learning: Participants underwent the community mental health consultation model program.
  Community mental health consultation model program : The community mental health consultation model program included collaboration among community mental health providers and (1) parent advocates to effectively maintain families in a school-based mental health program, (2) classroom teachers to enhance children's academic performance, and (3) peer-identified influential teachers to influence classroom teachers' use of behavior management strategies. This model further focuses on the strongest teacher and parent predictors of student learning.
Arm/Group | Links to Learning | Services as Usual
Number analyzed (Participants) | 100 | 65
units on a scale
  Baseline | 2.66 (.83) | 2.75 (.77)
  Spring Year 1 | 2.52 (.73) | 2.80 (.76)
  Fall Year 2 | 2.46 (.78) | 2.58 (.86)
  Spring Year 2 | 2.59 (.94) | 2.53 (.76)
  Fall Year 3 | 2.52 (.84) | 2.97 (1.05)
  Spring Year 3 | 2.62 (.81) | 2.79 (.79)

ADVERSE EVENTS:
Description: The study was not determined to present serious or non-serious adverse events to participants and therefore was given an expedited review by our Institutional Review Board (IRB). Thus, Serious and/or Other (non-serious) Adverse events were not collected or assessed.
Groups:
- Links to Learning: Participants will undergo the community mental health consultation model program.
  Community mental health consultation model program : The community mental health consultation model program includes collaboration among community mental health providers and (1) parent advocates to effectively maintain families in a school-based mental health program, (2) classroom teachers to enhance children's academic performance, and (3) peer-identified influential teachers to influence classroom teachers' use of behavior management strategies. This model further focuses on the strongest teacher and parent predictors of student learning.
- Services as Usual: Participants will receive treatment as usual and referrals.
  Treatment as usual (TAU) : TAU includes referral to community mental health clinic-based services, where participants will receive standard care for mental health-related problems.
Arm/Group | Links to Learning | Services as Usual
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was conducted in high poverty urban communities and therefore there were many impediments to recruitment and retention such as school closings and family migration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No